CLINICAL TRIAL: NCT02522455
Title: Flow-cycled Ventilation in Preterm Infants (FLIPI): A Pilot Study Looking at the Tolerance of Flow-cycled Ventilation by Preterm Infants With Respiratory Distress Syndrome
Brief Title: Flow-cycled Ventilation in Preterm Infants
Acronym: FLIPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R04003
Record Dates: First submitted 2015-08-09; First posted 2015-08-13 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Neonatal Respiratory Distress Syndrome
Keywords: Flow-cycled pressure-support ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preterm infants with RDS (Other)
  Interventions: Other: Flow-cycle ventilation; Other: Time-cycle ventilation mode

INTERVENTIONS:
Other: Flow-cycle ventilation — Pressure support level set as per previous pressure requirements to deliver a tidal volume of 5ml/kg (the same pressure amount used as the peak inspiratory pressure in the time-cycled mode)
  Other Names: Pressure-support ventilation
Other: Time-cycle ventilation mode — Peak inspiratory pressure set to deliver 5ml/kg tidal volume, Rate set as per previous requirements
  Other Names: Synchronised Intermittent Mandatory Ventilation

SUMMARY:
This short pilot study is to assess the tolerance of preterm infants, born below 32 weeks gestation with respiratory distress syndrome, to flow-cycle ventilation, and see if infants require less overall pressure from the ventilator than the usual conventional settings used, with the aim of providing data to construct a larger trial looking at the longer term outcome of these infants using this type of ventilation in the future.

Many preterm infants at these gestations require assistance from a ventilator due to the immaturity of their lungs. The lungs of preterm infants are susceptible to damage, especially if high pressures are needed or prolonged periods of ventilation. There is concern that if the infant's breathing pattern does not synchronise with the ventilator, this causes additional distress, longer duration of ventilation needed and increased risk of complications. Over the past 20 years, a different type of ventilation, known as flow-cycle ventilation, has been trialed, with limited use in preterm infants. This allows the baby to determine the duration of breathing in and out and how many breaths they require per minute. This would help babies to synchronise better with the ventilator, and consequently require less pressure from the ventilator.

This pilot study is being conducted at St. Mary's Hospital, Manchester. All babies born under 32 weeks gestation, with a stable respiratory effort, will be eligible for consideration for the study. The study will last no longer than 5 hours and involve the babies receiving different pressures from the ventilator in flow-cycle mode for 1-hour epochs. Blood gases after each epoch and continuous ventilator data will be downloaded to assess their tolerance on the different settings, before being returned to the usual conventional settings used on the unit. The babies will have continuous monitoring throughout as per standard neonatal intensive care.

DETAILED DESCRIPTION:
This study will be conducted as a short term, crossover study, where each infant will act as his or her own control and undertake all interventions within this study. The study is broken down into two parts in order to answer the two secondary research questions.

The limited studies looking at flow-cycled ventilation in preterm babies have been set up in a similar manner. Making each infant its own control limits the number of infants needed for this pilot study.

1. Prior preparations regarding protocol design

   The protocol has already been reviewed by the University of Leeds, by paper submission and viva to determine the suitability of the project from an educational point of view and suitability for the restricted time frame and resources available. Discussions with the neonatal unit technical support staff have already been undertaken to ensure that the study ventilators (an exact model to that used on the unit, but mobile) are configured with the required backup ventilation mode, to maintain the required level of breathing support, safety alarms and settings checked and the Eview box (device which allows the collection of data about the baby from the ventilator) installed as per manufacture guidelines.

   Training has also been given to the Principal investigator on the setup and maintenance of the study ventilator (the principal investigator is also a member of the clinical team who uses these ventilators on a daily basis and aware of how they are used).
2. Prior clinical care given & assessment for eligibility

   Prior to the study, eligible babies would have had a breathing tube inserted and surfactant medication given due to concerns with underdeveloped / immature lungs, fitting with being born at an early gestation. They would be receiving breathing support from the Engstrom Carestation Version 5.X (GE Healthcare) ventilator, the same ventilator used for the study, and would have received a dose of caffeine citrate intravenously to aid the infant's breathing drive, in line with unit policy and international consensus on managing respiratory distress syndrome in preterm infants. The clinical team may have deemed it necessary for monitoring and blood sampling to have inserted a catheter into one of the infant's arteries (an arterial line), though this is not a requisite for the study, but would be used for monitoring and sampling during the study if the infant was suitable. As per routine practice, the infants will have two methods of monitoring at all times. This would monitor oxygen saturations and heart rate as well as having monitoring on for blood pressure, breathing rate and temperature where deemed necessary.

   As both of the Principal and Chief Investigators are members of the clinical team on the neonatal intensive care unit at St. Mary's Hospital, it is easy to highlight suitable infants for the study from the patient lists and admissions to the unit, though prior discussion will take place with the attending neonatal team to discuss suitability. For any infant deemed potentially suitable after discussion with the attending clinical team, a parent information leaflet will be given to the parents at the time of greeting & introducing the study, after they have received an update on their baby's progress to date. As much time as possible will be allowed between this introduction and any attempt to answer questions and obtain written consent (minimum one hour) to allow the parents uncoerced thinking time.

   During this time, the research team will corroborate with the attending nurse / clinician and review the clinical data on the infant, including the x-rays done up until this time, the nursing observations and blood gas results, in order to assess for the inclusion and exclusion criteria. An eligibility form will be completed and signed by both a member of the research team and clinical team to ensure an agreement of eligibility. If there are concerns, the infant will not be recruited at this time.

   At an appropriate time for the parents, they will be approached by the Principal or Chief Investigator and any questions answered about the study. The research team will have to be happy that the parents have understood the information, implications, alternatives and are free to make a choice (as well as being eligible to consent legally). If the infant is suitable, a consent form will be completed. Randomisation will then occur by taking a sealed study envelope from the study box to find out which order they will undertake the different parts of the trial, and will be allocated a study number, which will be used on all documentation pertaining to the study, to ensure anonymity. (The study box would already have been pre-made with sealed envelopes containing information that has been generated from a random number database. The process of randomisation prevents there from being any influence on the final results purely due to the order in which the study parts are undertaken, making the study more robust to analyse. This has been a previous concern with other studies in the literature).

   The study ventilator (an exact model of the ventilator used on the unit) will be set up and safety checks undertaken, as well as the Eview box (the box which allows the ventilator data to be extracted and analysed though has no interference with the working of the ventilator itself) installed, safety back-up modes enabled to ensure that the infant has sufficient breathing support from the ventilator in the event that they do not maintain a strong breathing pattern, and the study number and weight of the child be accurately entered into the ventilator by the research team.

   The researcher will then examine the infant to ensure that the time of commencing the study the infant still satisfies the criteria for inclusion and is deemed 'stable' and a blood gas sample will be taken from the baby (either from the pre-sited arterial line if available or from the capillaries in the foot according to standard practice; distress and amount of blood will be minimised and should not cause any instability). This sample will be analysed by the machines routinely used on the intensive care unit, and any other blood tests that the infant may need (e.g. blood sugar monitoring, which is usually done every 2-4 hours at this stage) will be performed at the same time / on the same sample of blood (if possible) to minimise distress and interventions. A special nursing observation chart will be commenced at this time by the attending nurse / research team, recording the routine observations that any ventilated infant would require. This first set of observations (on the pre-study ventilator settings) would be the baseline settings, allowing any deviation from this stability to be highlighted and acted upon early.
3. First part of study

   The infant would be switched onto the study ventilator, a process which takes less than a second, and involves disconnecting the old ventilator tubing from the breathing tube reconnecting it to the new ventilator tubing. This is necessary in order for Eview box to work (the original ventilator would have to be turned off for a short period of time, which would not be ethical to leave the baby without controlled breathing support). Care would be taken not to dislodge the breathing tube whilst the infant was examined to ensure that the chest was rising and that the ventilator was receiving data from the infant. The time on the ventilator would be noted down on the observation chart to aid with data analysis later.

   Depending on randomisation, the infant would either receive a high pressure or low pressure from the study ventilator.
   * All other settings would match those that the infant was on beforehand where possible. (The high and low pressures are pre-set based on what pressure the infant was requiring before the study with either 80% of this (low pressure) or 120% of this (high pressure) these limits are deemed to be safe and within acceptable clinical practice).
   * The infant would remain on this setting for 1 hour.
   * Their nursing observations will be recorded every 15 minutes, including a blood pressure if they did not have an arterial line to read it continuously (this is not unusual practice as the baby would receive this intensity of observation if they were having a blood transfusion).

   After the end of the hour, a blood gas would be taken, and the ventilator would be switched to the other setting (either low pressure, if the infant previously received high pressure, or vice versa). The same process would be repeated in terms of the timings and observations taken. The time on the ventilator would be noted for analysis purposes when the pressures were switched.

   After the second hour, the blood gas would be repeated and the infant placed back on the initial ventilator, on a setting appropriate for the condition of the infant at that time. This completes the first part of the study and the infant would resumed routine care for a least an hour. A blood gas would be taken after 1 hour as per usual convention to ensure that they are stable and settled back onto the initial ventilator.
4. Second part of the study

   After 1 hour back on the standard ventilator, the infant would be reassessed to ensure that they were stable. If this is the case, as stated above, a blood gas would be taken and part two of the study commenced. The observations recorded would provide a baseline for the second part of the study. The infant would once again be switched back to the study ventilator and time noted.

   Depending on the initial randomisation, the infant would either receive time-cycled ventilation (the usual convention) or flow-cycled ventilation (as in part one of the study) from the study ventilator.
   * All other settings would match those that the infant was on beforehand where possible.
   * The infant would remain on this setting for 1 hour.
   * Their nursing observations will be recorded every 15 minutes, including a blood pressure if they did not have an arterial line to read it continuously.

   After the end of the hour, a blood gas would be taken, and the ventilator would be switched to the other setting (either flow-cycled, if the infant previously received time-cycled, or vice versa). The same process would be repeated in terms of the timings and observations taken.

   The time on the ventilator would be noted for analysis purposes when the pressures were switched.

   After the second hour, the blood gas would be repeated and the infant placed back on the initial ventilator, on a setting appropriate for the condition of the infant at that time. This completes the second and final part of the study and the infant would resume routine care for the duration of their stay on the unit. A blood gas would be taken after 1 hour as per usual convention to ensure that they are stable and settled back onto the initial ventilator.
5. After completion of study

   After the study had been completed, there would be a handover of care back to the attending clinical team with update to the clinical team and parents (if present) regarding the clinical condition of the baby.

   Regarding the data, the encrypted flash disk will be removed from the study ventilator and the data downloaded on an NHS computer on the unit. This data, along with the nursing observation charts and blood gas results, will then be reviewed by the independent consultant neonatologist for safety and quality assurance prior to a second baby undergoing the study.

   The researcher is responsible for ensuring that the study ventilator is cleaned appropriately in line with the manufactures and unit guidelines and is ready for any future participants.
6. Safety interventions

These have been highlighted in the main issues question where there is a break from protocol due to safety concerns. It is clear in the protocol what needs to be done if there are concerns. Only one baby will undergo the study at any one time and any concerns will be reviewed by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 32 weeks gestation at time of study enrolment
* Evidence of Respiratory Distress Syndrome (Clinical signs of respiratory distress, need for surfactant / ventilation, any O2 requirement with typical Chest radiograph appearance)
* Patients to have received loading dose of caffeine, as per unit policy
* Informed parental consent given
* Intubated and requiring continuing ventilatory support
* Exogenous surfactant given if indicated (6 hours or more before study entry)
* Cardiovascular status stable for at least 3 hours before study
* Stable on ventilation with satisfactory blood gases & inspired oxygen concentration < 40% at time of starting study, and for the preceding 3 hours
* Regular spontaneous respiratory effort, consistently triggering the ventilator in SIMV mode, for at least 3 hours prior to the start of the study
* Less than 24 hours of age at the start of the study

Exclusion Criteria:

* Refusal or withdrawal of parental consent
* Major congenital abnormality, including any need for surgery
* Known large intracranial haemorrhage (grade 3 or 4 intraventricular haemorrhage or other significant intracranial abnormality)
* Seizures
* Pneumothorax or pulmonary interstitial emphysema
* Inspired oxygen requirement > 40% after surfactant administration

Ages: 6 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mean airway pressure used | 6 hours
  Amount of pressure required in either ventilation mode
Inspiratory time | 6 hours
  Amount of time the infant require inspiratory support from the ventilator (in flow-cycle mode only)
Respiratory rate | 6 hours
  Spontaneous respiratory rate from infant in either ventilation mode

SECONDARY OUTCOMES:
Exhaled tidal volume | 6 hours
  Amount of gas exhaled (measured in mls, ml/kg body weight)
Exhaled minute ventilation | 6 hours
  Product of exhaled tidal volume and respiratory rate
Oxygen requirement | 6 hours
Acid - base balance | In each 1-hour epoch (end of)
  Assessment of pH and carbon dioxide clearance in each ventilation mode

OTHER OUTCOMES:
Rapid shallow breathing index | 6 hours
  Measure of respiratory effort required by infant: calculated by respiratory rate divided by exhaled tidal volume

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Mitchell, MD FRCPCH, Study Director — Manchester University NHS Foundation Trust
Locations (1):
- St. Mary's Hospital, Manchester, United Kingdom

REFERENCES:
- [Background] Attar MA, Donn SM. Mechanisms of ventilator-induced lung injury in premature infants. Semin Neonatol. 2002 Oct;7(5):353-60. doi: 10.1053/siny.2002.0129. PMID 12464497
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Donn SM, Sinha SK. Minimising ventilator induced lung injury in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F226-30. doi: 10.1136/adc.2005.082271. PMID 16632652
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Halliday HL; European Association of Perinatal Medicine. European consensus guidelines on the management of neonatal respiratory distress syndrome in preterm infants--2013 update. Neonatology. 2013;103(4):353-68. doi: 10.1159/000349928. Epub 2013 May 31. PMID 23736015
- [Background] Kapasi M, Fujino Y, Kirmse M, Catlin EA, Kacmarek RM. Effort and work of breathing in neonates during assisted patient-triggered ventilation. Pediatr Crit Care Med. 2001 Jan;2(1):9-16. doi: 10.1097/00130478-200101000-00003. PMID 12797881
- [Background] Schulzke SM, Pillow J, Ewald B, Patole SK. Flow-cycled versus time-cycled synchronized ventilation for neonates. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD008246. doi: 10.1002/14651858.CD008246.pub2. PMID 20614468
- [Background] Jarreau PH, Moriette G, Mussat P, Mariette C, Mohanna A, Harf A, Lorino H. Patient-triggered ventilation decreases the work of breathing in neonates. Am J Respir Crit Care Med. 1996 Mar;153(3):1176-81. doi: 10.1164/ajrccm.153.3.8630564.
- [Background] Schmalisch G, Wilitzki S, Wauer RR. Differences in tidal breathing between infants with chronic lung diseases and healthy controls. BMC Pediatr. 2005 Sep 8;5:36. doi: 10.1186/1471-2431-5-36. PMID 16150146
- [Background] Abd El-Moneim ES, Fuerste HO, Krueger M, Elmagd AA, Brandis M, Schulte-Moenting J, Hentschel R. Pressure support ventilation combined with volume guarantee versus synchronized intermittent mandatory ventilation: a pilot crossover trial in premature infants in their weaning phase. Pediatr Crit Care Med. 2005 May;6(3):286-92. doi: 10.1097/01.PCC.0000161071.47031.61. PMID 15857526
- [Background] De Luca D, Conti G, Piastra M, Paolillo PM. Flow-cycled versus time-cycled sIPPV in preterm babies with RDS: a breath-to-breath randomised cross-over trial. Arch Dis Child Fetal Neonatal Ed. 2009 Nov;94(6):F397-401. doi: 10.1136/adc.2009.162446. Epub 2009 Jul 1. PMID 19574255
- [Background] Gupta S, Sinha SK, Donn SM. The effect of two levels of pressure support ventilation on tidal volume delivery and minute ventilation in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2009 Mar;94(2):F80-3. doi: 10.1136/adc.2007.123679. Epub 2008 Aug 1. PMID 18676412
- [Background] Osorio W, Claure N, D'Ugard C, Athavale K, Bancalari E. Effects of pressure support during an acute reduction of synchronized intermittent mandatory ventilation in preterm infants. J Perinatol. 2005 Jun;25(6):412-6. doi: 10.1038/sj.jp.7211303. PMID 15843812